CLINICAL TRIAL: NCT03209921
Title: Pharmacokinetic Variability of Daptomycin During Prolonged Therapy for Bone and Joint Infections
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0464
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Bone and Joint Infection; Patient Treated by Daptomycin
Keywords: Bone and Joint Infection; Daptomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Daptomycin is a cyclic lipopeptide that has been proposed as an alternative therapeutic option in patients with prosthetic joint infection caused by Staphylococcus or Enterococcus species in the latest Infectious Diseases Society of America (IDSA) guidelines.

The population pharmacokinetics (PK) of daptomycin have been described in various groups of patients in previous publications. However, little information exists on the PK of daptomycin in patients with bone and joint infections (BJI). Also, previous population studies did not investigate daptomycin PK over prolonged therapy, and, to our knowledge, no study has reported the intraindividual PK variability of this drug.

The aim of this study is to describe the inter- and intraindividual PK variability of this drug.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with daptomycin for BJI in Lyon Center in 2012 and 2013

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with daptomycin for BJI in Lyon Center in 2012 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Typical daptomycin clearance | 6 months
  Mean daptomycin plasma clearance (unit, liters per hour)
  Outcome measures performed regularly in those patients throughout therapy, roughly every month.
Typical daptomycin volume of distribution | 6 months
  Mean daptomycin volume of distribution (unit, liters) in the population